CLINICAL TRIAL: NCT02660697
Title: 3D Radiographic Evaluation of Post-extraction Healing Following Treatment With a Novel Implant Site Development Technique
Brief Title: 3D Radiographic Evaluation of a Novel Implant Site Development Technique
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Balint Molnar, Dr. Balint Molnar DMD, PhD, assistant professor, Semmelweis University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XSD-Semmelweis-Perio
Record Dates: First submitted 2016-01-18; First posted 2016-01-21 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Tooth Extraction Status Nos; Edentulous Alveolar Ridge
Keywords: socket preservation, implant site development

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Test - Extraction site development group (Active Comparator): In the test group 29 healthy patients presenting 33 single rooted teeth scheduled for extraction with Extraction Defect Sounding (EDS) Class 3-4 type buccal bony dehiscences were included. 29 maxillary single rooted teeth and 4 single rooted teeth in the mandible (27 incisors, 2 canines and 4 premolars) were removed and treated by the novel extraction site development method. Pre- and postoperative ConeBeam Computer Tomography (CBCT) data were collected for further analysis.
  Interventions: Procedure: Extraction site development
- Control - Spontaneous healing group (No Intervention): In the control group. pre- and postextraction CBCT data sets of 14 patients with 21 extracted teeth were collected. 11 maxillary single rooted teeth and 10 single rooted teeth in the mandible (13 incisors, 2 canines and 6 premolars) were extracted and left for spontaneous healing.

INTERVENTIONS:
Procedure: Extraction site development — In the test group, extraction sockets presenting EDS Type 3-4 buccal bony dehiscences were treated by a novel minimally invasive tunnelised modified GBR approach (XSD).
  Other Names: XSD
  Arms: Test - Extraction site development group

SUMMARY:
The present retrospective study aims at assessing the clinical effects of a novel implant site development (Extraction site development - XSD) technique after tooth extraction compared with extraction alone in patients requiring dental implant placement following healing of extraction sockets.

DETAILED DESCRIPTION:
In advanced (Extraction Defect Sounding Class 3-4) alveolar defects, a minimally invasive tunnelised socket preservation technique utilising long term resorbable membranes and connective tissue grafting was used for extraction site development (XSD). The novel technique was evaluated in a retrospective comparative case series study including a total of 54 extraction sites. In the test group, out of 33 single rooted teeth, 29 in the maxilla and 4 in the mandible were removed, extractions sites were treated by the XSD method. Out of 33 teeth, 27 were incisors, 2 canines and 4 premolars. In the control group, out of 21 single rooted teeth, 11 in the maxilla and 10 in the mandible were extracted and left for spontaneous healing. Out of 21 teeth, 13 were incisors, 2 canines and 6 premolars. CBCT scans were taken prior to tooth extraction and 6-9 months later in both groups. Radiographic evaluation was carried out using the I-CAT Vision (Imaging Sciences International, LLC; Hatfield, USA) and ImageJ (National Institutes of Health) softwares. Following manual alignment of CBCTs vertical and horizontal linear measurements as well as planimetric measurements of cross-section areas were performed in pre- and postoperative data sets at the extraction sites.

ELIGIBILITY:
Inclusion Criteria:

Presence of at least 1 single rooted tooth scheduled for extraction with EDS Class 3-4 type buccal bony dehiscence

Exclusion Criteria:

Exclusion criteria int he test group included uncontrolled inflammation at the surgical site, full mouth plaque or bleeding scores more than 20%, diabetes, pregnancy, known metabolic bone diseases, smoking more than 10 cigarettes a day, history of any relevant systemic diseases, radiotherapy chronic use of bisphosphonates or systemic steroids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2007-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Orovestibular socket dimension | From baseline to 6-9 months postoperatively
  On prealigned pre- and postoperative CBCT cross-sections, linear measurements were taken parallel to a reference base to determine the orovestibular width of extractions sites

SECONDARY OUTCOMES:
Minimal orovestibular socket dimension feasible for implant placement | From baseline to 6-9 months postoperatively
  Minimal orovestibular socket dimension feasible for implant placement was defined as 6mm
Vertical socket dimension | From baseline to 6-9 months postoperatively
  On prealigned pre- and postoperative CBCT cross-sections, linear measurements were taken perpendicularly to a reference base to determine the height of extractions sites
Socket area | From baseline to 6-9 months postoperatively
  On prealigned pre- and postoperative CBCT cross-sections, planimetric measurements were taken to determine the cross-section area of extractions sites

CONTACTS AND LOCATIONS:
Overall Officials: Balint Molnar, DMD, PhD, Principal Investigator — Semmelweis University Department of Periodontology
Locations (1):
- Semmelweis University Department of Periodontology, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No